CLINICAL TRIAL: NCT06861868
Title: Early Brain Development and Child Nutrition and Obesity
Brief Title: Brain and Behavior Influences on Obesity Development From Infancy Through Childhood
Acronym: RESONATE
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Rhode Island Hospital (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00118376; R01DK136602 (NIH)
Record Dates: First submitted 2025-02-12; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Overweight
Keywords: obesity; overweight; pediatric; eating behavior; appetite; neuroimaging; magnetic resonance imaging; brain development
MeSH Terms: conditions — Obesity; Overweight; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators project, RESONATE, aims to investigate why some children develop obesity. To do this it uses data on eating and eating-related behaviors, genetic and environmental factors, and brain structure and function. This data is collected in a sub-sample of RESONANCE, a large study of families of children from infancy through childhood. The results will lay foundations for the development of early interventions to prevent or treat obesity.

DETAILED DESCRIPTION:
Obesity risk shows individual variation such that some children are more likely than others to gain excess weight. One potential reason is that, due to genetic and environmental factors, individuals vary in appetitive behaviors that drive food intake and weight. However, the neurodevelopmental mechanisms underpinning variation in appetite and weight, and effects of risk and protective factors on those outcomes, are not understood. Preliminary data from RESONANCE, the investigators large MRI cohort, suggests obesity risk factors such as maternal pre-pregnancy obesity and obesity-associated genetic variants are associated with not just heightened parent-reported child appetite and adiposity, but with altered patterns of brain structure development from infancy through early childhood. However the relevance of these findings to appetitive behaviors and development of obesity in middle childhood is unknown. This is important because obesity rates and metabolic complications increase through development, adiposity and eating habits measured in later childhood track into adulthood, and obesity is harder to treat later in development, making middle childhood a key stage for capturing outcomes with relevance for lifetime metabolic health. Further, although functional magnetic resonance imaging (MRI) studies have identified altered patterns of activation in brain appetite circuits in association with pediatric obesity and early risk factors for obesity, the predictors of altered functioning of brain appetite circuits in middle childhood are unknown. Identifying the patterns of brain development that predict obesity-promoting behaviors and brain functioning in middle childhood is essential to understand the neural mechanisms by which early obesity risk factors drive excess intake and obesity, and may help pinpoint neurobehavioral targets for early obesity prevention. Finally, although preclinical research and MRI studies of children under 9 years of age support that hypothalamic gliosis, a cellular inflammatory response, plays a role in obesity pathogenesis, it is unclear whether it occurs or impacts appetite in earlier life. For the proposed study, RESONATE, the investigators will address the above research gaps by extending the RESONANCE study to administer meal tests, behavioral and functional magnetic resonance imaging (fMRI) tasks assessing food and non-food reward and cognitive control, and weight/ adiposity measures in middle childhood, and examining hypothalamic gliosis, in a sub-sample of RESONANCE children. By combining this data with extant MRI data and extant or newly-collected data on obesity risk and protective factors, the investigators will test a multi-faceted hypothesis that prenatal, genetic and postnatal factors lead to differential early development of brain appetite circuits, which in turn gives rise to variation in appetitive behaviors and behaviors involving reward processing and cognitive control as well as altered function of brain appetite circuits, that act to influence the development of obesity into middle childhood. The investigator's long-term goal is to lay foundations for developmentally-appropriate, neurobehaviorally-informed interventions to address child obesity.

ELIGIBILITY:
Inclusion Criteria:

* Participants from the RESONANCE cohort are eligible if the participant will reach 7-12 years of age during the proposed project period and have no food allergies.

Exclusion Criteria:

* Exclusion criteria for RESONANCE include:

  1. In utero exposure to alcohol, cigarette, or illicit substances;
  2. First trimester fetal US abnormalities;
  3. Complicated pregnancy (e.g., pre-eclampsia);
  4. Complicated delivery, including APGAR scores less than 8 and/or neonatal intensive care unit (NICU) admission;
  5. History of neurological (e.g., epilepsy), psychiatric (e.g., anxiety or depression requiring treatment with medication) or developmental disorder (e.g., autism spectrum disorder (ASD), dyslexia);
  6. Contraindications for MRI including metal in the body, claustrophobia.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are drawn from the existing RESONANCE cohort. RESONANCE is a large community sample of families of children ranging from infancy through middle childhood.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Meal test intake as assessed by total kilocalories consumed | Day 1
  Total kilocalories consumed. Once at the first study visit (lab visit)
Weight/adiposity as assessed by BMI | Day 1
  Body Mass Index z-score. Once at the first study visit (lab visit)
Food-related reward as assessed by food-related delay discounting task | Day 1
  Number of trials the child passes. Once, at the first study visit (lab visit)
Food-related cognitive control as assessed by food-related go/no-go task | Day 1
  Commission error rate. Once, at the first study visit (lab visit)
Functioning in brain appetite circuits as assessed by cue reactivity task | During MRI procedure
  Activation of striatal reward regions and fronto-cingulate control circuits during task assessing food-related reward (cue reactivity). Once, at the second study visit (MRI visit).
Functioning in brain appetite circuits as assessed by cognitive control task | During MRI procedure
  Activation of striatal reward regions and fronto-cingulate control circuits during task assessing food-related cognitive control (go/no go). Once, at the second study visit (MRI visit).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Carnell, PhD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Hugo W. Moser Research Institute at Kennedy Krieger, Inc., Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
RESONATE is a sub-study within a sub-sample drawn from the RESONANCE cohort, supported by NIH's ECHO initiative. RESONANCE data used for RESONATE will include data on anthropometrics, parent-report appetitive behaviors, executive functioning, child diet, food parenting, maternal pre-pregnancy body weight, sociodemographic characteristics, common genetic variants, and brain MRI measures. For RESONATE, additional data including behavioral task responses, data from eating behavior tests, structural and functional brain MRI measures, and survey responses including measures of eating-disordered behaviors and food parenting, will be obtained in children assessed age 7-12 years. All RESONANCE data collected under the ECHO-wide protocol will be made publicly available via the National Institute of Child Health and Human Development Data and Specimen Hub. Data unique to the RESONATE sub-study will also be preserved and made available for sharing on request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: RESONANCE data collected as part of the wider ECHO study is uploaded to ECHO's central databases on a regular basis and will be made available to the public after regular periodic datalocks as determined by the ECHO program. RESONATE data will be made available at the time of publication of those data and will be available for a minimum of five years after any publication on which it is based.
Access Criteria: Data from RESONATE and RESONANCE will be available for investigators providing an Institutional Review Board (IRB)/Ethics approval or certification of exemption from IRB/Ethics review, and agreeing to the terms and conditions of a data use agreement. Data will be available for any purpose unless prohibited by the informed consent process. To request access to RESONANCE data collected as part of the wider ECHO study, researchers will request a DASH account and submit a Data Request Form. The NICHD DASH Data Access Committee will review the request and provide a response in approximately two to three weeks. Once granted access, researchers will be able to use the data for three years. RESONATE data can be requested from the PIs and will be reviewed on a rolling basis. To protect participants, the investigators will deidentify shared data to the greatest extent possible, using masked study identifiers and utilizing HIPAA-compliant procedures.